CLINICAL TRIAL: NCT04797585
Title: A Prospective Randomized Trial Comparing Vaginal Hysterectomy and Laparoscopic Supracervical Hysterectomy at the Time of Sacrocolpopexy for the Treatment of Uterovaginal Prolapse
Brief Title: Vaginal Hysterectomy vs Supracervical Hysterectomy at the Time of Sacrocolpopexy
Acronym: ColoplastLSC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-1293
Record Dates: First submitted 2021-03-10; First posted 2021-03-15 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Vaginal Hysterectomy; Laparoscopic Supracervical Hysterectomy
MeSH Terms: interventions — Hysterectomy, Vaginal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic supracervical hysterectomy (Active Comparator): Minimally invasive procedure to remove a woman's uterus
  Interventions: Other: Laparoscopic supracervical hysterectomy
- Vaginal hysterectomy (Experimental): Surgical procedure to remove the uterus
  Interventions: Other: Vaginal hysterectomy

INTERVENTIONS:
Other: Laparoscopic supracervical hysterectomy — Laparoscopic supracervical hysterectomy
  Arms: Laparoscopic supracervical hysterectomy
Other: Vaginal hysterectomy — Vaginal hysterectomy
  Arms: Vaginal hysterectomy

SUMMARY:
The primary objective of the proposed study is to determine the difference in surgical time between minimally invasive (laparoscopic) sacrocolpopexy performed with concurrent vaginal hysterectomy versus laparoscopic supracervical hysterectomy. The secondary objectives are to determine if there are differences in intraoperative adverse events and postoperative mesh-related complications and prolapse recurrence between the groups.

DETAILED DESCRIPTION:
Study Procedures:

Study Identification and Recruitment Potential subjects will be identified by members of the Center for Urogynecology & Pelvic Reconstructive Surgery at the Cleveland Clinic Main campus, Hillcrest Hospital and Fairview Hospital. Eligible patients who agree to participate will be provided written informed consent administered by the collaborators listed on this IRB.

Randomization All subjects will be predetermined by their surgeon to undergo a laparoscopic sacrocolpopexy. The participants will then be randomized to either concurrent vaginal hysterectomy or laparoscopic supracervical hysterectomy according to a computer-generated randomization schedule with the use of the SAS statistical software package (SAS Institute, Cary, NC).

Office Interventions All patients will be seen for a preoperative visit and then postoperatively at 6, 12 and 24 months. The 6 month visit will be standard of care, the 12 month and 24 month visit will be a research visit. At each visit, a vaginal exam and a complete Pelvic Organ Prolapse Quantification (POP-Q) exam will be performed. In addition, patients will be asked to complete the Pelvic Floor Distress Inventory (PFDI-20), Incontinence Severity Index (ISI), Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12) and Patient Global Impression of Improvement (PGII) questionnaires at the pre-operative visit as well as the 6, 12, and 24 month postoperative visits. Completion of these questionnaires is the only additional assessment that is specific to participation in this study and is not usually included as part of the standard care of sacrocolpopexy. It should take no more than 10-15 minutes to complete the questionnaires. The study subjects will not be exposed to any additional risk by participating in this study except for the inconvenience of completing the questionnaires.

Surgical Interventions The laparoscopic portions of the surgery will be performed using four ports: an umbilical port for the laparoscope (either 5 or 10/12mm), two ports (either 5, 8 or 10/12 mm) in the bilateral lower quadrants, and one 5-mm port placed at the level of the umbilicus, lateral to the rectus muscle on either side for retraction.

If a supracervical hysterectomy is to be performed, it will be done in a standard fashion. A uterine manipulator will be placed inside of the uterus. The round ligaments will be transected using cautery. The fallopian tubes and ovaries will be left in situ or removed at the time of hysterectomy depending upon the preoperative decision made between the surgeon and patient. The uterine arteries and cardinal ligaments will be cauterized laparoscopically. The uterus will be amputated at the level of the internal cervical os and the endocervical canal will be cauterized. The specimen will be extracted in a laparoscopic endocatch bag and removed through an extended incision at the umbilicus at the end of the case. Dissection of the vagina anteriorly and posteriorly will be done laparoscopically with the use of an end-to-end anastomosis (EEA) sizer in the vagina. Dissection of the presacral space will also be done laparoscopically. Five to six 2-0 PDS sutures will be placed to secure the mesh to the anterior vagina as well as the posterior vagina for a total of 10-12 sutures on the vagina; the arm of the mesh will be secured to the anterior longitudinal ligament of the sacrum using two 0 Prolene sutures. The Coloplast® Restorelle Y mesh will be used for all cases. The peritoneum will be closed with 0 or 2-0 vicryl sutures.

If a vaginal hysterectomy is performed, it will be done in a standard fashion using a traditional clamp and suture technique starting at the uterosacral ligaments and ending with the utero-ovarian ligaments. The specimen will be extracted through the vagina. Dissection of the vagina anteriorly and posteriorly will be done vaginally. The mesh will be attached vaginally using five to six 2-0 PDS sutures on the anterior and posterior vagina for a total of 10-12 sutures on the vagina. The Coloplast® Restorelle Dual flat mesh will be used. The vagina will then be closed in two layers using 0 or 2-0 vicryl suture. Laparoscopic entrance will then be gained and set up will be done as described above. The presacral space will be dissected laparoscopically and the mesh attached to the anterior longitudinal ligament of the sacrum using two 0 Prolene sutures. The peritoneum will be closed with 0 or 2-0 vicryl sutures.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18, who are to undergo laparoscopic sacrocolpopexy for uterovaginal prolapse and desire concurrent hysterectomy at the time of surgery
* Other concomitant laparoscopic or prolapse and anti-incontinence procedures (cystocele repair, rectocele repair or mid-urethral sling procedures) will be performed at the primary surgeon's discretion.
* Patient's must have an up-to-date PAP smear on record, or a PAP smear is performed in the office and verified to be normal pre-enrollment

Exclusion Criteria:

* Inability to comprehend written and/or spoken English
* Inability to provide informed consent
* Medical illness precluding laparoscopy
* Need for concomitant surgeries not related to pelvic organ prolapse or incontinence
* Sacrocolpoperineopexy
* Patients desiring uterine preservation (hysteropexy)
* Previous apical prolapse surgery (hysteropexy)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women undergoing hysterectomy
Enrollment: 3 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2023-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cecile Ferrando, M.D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nassif J, Yadav GS, Orejuela FJ, Turrentine MA. Rate of Mesh Erosion After Sacrocolpopexy With Concurrent Supracervical Compared With Total Hysterectomy: A Systematic Review and Meta-analysis. Obstet Gynecol. 2022 Sep 1;140(3):412-420. doi: 10.1097/AOG.0000000000004901. Epub 2022 Aug 3. PMID 35926201

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Laparoscopic Supracervical Hysterectomy | Vaginal Hysterectomy
Started | 1 | 2
Completed | 1 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Laparoscopic Supracervical Hysterectomy | Vaginal Hysterectomy | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 1 | 2 | 3
Age, Continuous [Mean (Full Range); unit: Years] | NA [68 to 68] — Measure of dispersion n/a as only one participant. | 70.5 [70 to 71] | 69.7 [68 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 2 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Total Surgical Time - Time of Incision to Time of Sacrocolpopexy Completion
Description: Completion = time of abdominal incisions closed
Time Frame: One day intraoperative
Measure: Mean (Full Range); unit: Minutes
Arm/Group | Laparoscopic Supracervical Hysterectomy | Vaginal Hysterectomy
Number analyzed (Participants) | 1 | 2
Minutes | NA [253 to 253] — Measure of central tendency is n/a as there is only one participant. | 387.5 [379 to 396]

2. Secondary Outcome: Post-operative Mean Difference PFDI-20 at 24 Months
Description: Mean difference between baseline (pre-operative) and 24 months post-procedure. The Pelvic Floor Disability Index (PFDI-20) is a is a short form that gives a comprehensive assessment of the effect of pelvic floor disorders. The scale exists from 0-4 (0=not present, 4=quite a bit)
Time Frame: 24 months
Reporting Status: Not Posted

3. Secondary Outcome: Post-operative Mean Difference ISI at 24 Months
Description: Mean difference between baseline (pre-operative) and 24 months post-procedure. The Incontinence Severity Index (ISI) consists of two questions, regarding frequency and amount of leakage. It categorizes urinary incontinence (UI) into slight, moderate, severe, and very severe. The scale exists from 0-12 (0=none, 12=very severe).
Time Frame: 24 months
Reporting Status: Not Posted

4. Secondary Outcome: Post-operative Mean Difference PGII at 24 Months
Description: Mean difference between baseline (pre-operative) and 24 months post-procedure. The Patient Global Improvement Indices (PGII) is a seven-item measure which measures symptoms and degree of bother. The scale exists from 0-7 (0=very much better, 7=very much worse).
Time Frame: 24 months
Reporting Status: Not Posted

5. Secondary Outcome: Post-operative Mean Difference PISQ-12 at 24 Months
Description: Mean difference between baseline (pre-operative) and 24 months post-procedure. The Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12) is a validated and reliable short form that evaluates sexual function in women with urinary incontinence and/or pelvic organ prolapse. The scale exists from 0-4 (0=never, 4=always).
Time Frame: 24 months
Reporting Status: Not Posted

6. Secondary Outcome: Postoperative Subjective Recurrence at 24 Months
Description: Subjective recurrence is defined as patients who complain of vaginal bulge sumptoms (Question #3 on the PFDI-20)
Time Frame: 24 months
Reporting Status: Not Posted

7. Secondary Outcome: Reported Mesh Erosion at 24 Months
Description: Mesh erosion is defined as presence of eroded mesh in the vagina on examination postoperatively up to 24 months after surgery
Time Frame: 24 months
Reporting Status: Not Posted

8. Secondary Outcome: Postoperative Objective Recurrence at 24 Months
Description: Objective recurrence is defined by POP-Q: Apical descent greater than one-third of total vaginal length or anterior or posterior vaginal wall beyond the hymen
Time Frame: 24 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 Months
Arm/Group | Laparoscopic Supracervical Hysterectomy | Vaginal Hysterectomy
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 0/1 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-30): https://cdn.clinicaltrials.gov/large-docs/85/NCT04797585/Prot_SAP_000.pdf
  • Informed Consent Form (2022-08-10): https://cdn.clinicaltrials.gov/large-docs/85/NCT04797585/ICF_001.pdf